CLINICAL TRIAL: NCT03229824
Title: Randomized Controlled Trial to Reduce Surgical Site Infections in Breast Cancer Surgery With Clorhexidine Gluconate Securement Dressing (Tegaderm CHG)
Brief Title: Use of Clorhexidine Dressings to Reduce Surgical Site Infections in Breast Cancer Surgery. A Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, MYRNA CANDELARIA, MD PHD, Ethics Commissioner, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEI/1090/16
Record Dates: First submitted 2017-04-21; First posted 2017-07-26 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Drain antisepsis; Bacterial colonization; Surgical site infection
MeSH Terms: conditions — Breast Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiseptic occlusive dressing group (Experimental): A chlorhexidine gluconate occlusive adhesive dressing (Tegaderm CHG) will be applied to the intervention drain sites and changed every seven days.
  Interventions: Device: Antiseptic occlusive dressing group
- Standard care (No Intervention): Standard drain care will be performed twice a day or three times if bulb is full and needs to be emptied. Standard drain care consists of stripping the tubing, emptying the drainage bulb, recording the volume of fluid, and cleaning the drain site and the tubing with a cotton swab dipped in rubbing alcohol.

INTERVENTIONS:
Device: Antiseptic occlusive dressing group — A chlorhexidine gluconate occlusive adhesive dressing (Tegaderm CHG) will be applied to the intervention drain sites and changed every seven days.
  Other Names: Tegaderm CHG Dressing
  Arms: Antiseptic occlusive dressing group

SUMMARY:
Surgical site infection (SSI) after breast and axillary surgery occurs more often than for other clean surgical procedures. Infection in the setting of sick woman could delay the adjuvant therapy and result increase morbidity and mortality. Also this increased costs associated with health care.Surgical drains have been noted as a potential source for surgical site infections. The primary aim of the study is to determine if chlorhexidine occlusive dressings applied to the intervention drain sites effectively decreases rates of bacterial colonization in drain fluid and drain tips compared to standard care.

DETAILED DESCRIPTION:
Following approval by the National Cancer Institute Review Board, eligible subjects will be recruited prospectively from the Breast Cancer Department at National Cancer Institute, México from November 2016 to November 2017. Individuals with confirmed cancer undergoing total mastectomy (TM), modified radical mastectomy (MRM) and/or axillary lymph node dissection (ALND) in which surgical drains are going to be used will be identified through the surgical scheduling sheet. If the subjects are eligible according to the inclusion criteria, the will be interviewed by one of the main researchers. In the initial interview the informed consent will be read and signed. Also the study coordinator will collect the data of interest from the medical records and will register it in a data collection sheet specially created for this project.

Following informed consent, participants will be randomize to either the standard drain care regimen or the drain antisepsis regimen by a computerized randomization program, using dynamic allocation and stratifying by surgical procedure (radical surgery or conservative surgery). Subjects who had bilateral cancer underwent to the same regimen for both sides. The operating surgeon will know the assigned treatment arm at the end of the surgery.

The surgery will consist on placing a chlorhexidine gluconate occlusive adhesive dressing to the drains side at the end of the surgery. The dressing will be changed each 7 (+-1) days until the drain is removed.

All the participants and the principal take-carers, despite of the group of participation, will be personal instructed by a member of the research team in the first hours of the postoperative, before the departure. In addition, they will be given paper based instructions for the general care of the drain and the surgery wound.

For the experimental group, the dressing will be changed each 7(+-1) days; The site of the insertion must be cleaned with 70% concentration isopropyl alcohol towels. The evaluation and quantification of the drained fluid will be done every 12 hours as it is done usually in these patients.

The patients will be followed for 30 days from the surgery until the resolution of the infectious complication, if it occurs. The patients will go at the end of the first postoperative week (POP 7+-1). In each visit, the coordinator of the study will register the information of the patient in the register sheet. In each visit the patient will be evaluated, the characteristics of the surgical wound and the characteristics of drain fluid will be consigned in the protocol register sheet. The investigator will verify that the participants have correctly done the clean-up the drain.

All patients will undergo semiquantitative cultures of the drain bulb at the first and second week postoperative. Also the investigators will take the distal part of the internal segment of each removed drainage tube for semiquantitative culture. All participants will be evaluated for clinical signs of infection and for any adverse reactions to the drain antisepsis at the follow-up visits. In case of a surgical site infection, the patient will receive the right treatment and will remain in surveillance until the resolution.

ELIGIBILITY:
Inclusion Criteria:

* Females minimum age 18 able to give informed consent
* Breast cancer confirmed by histopathology
* Patients undergoing unilateral or bilateral mastectomy with or without immediate expander reconstruction.

Exclusion Criteria:

* Males
* Patients who deny informed consent
* Prior radiation therapy to the sick breast.
* Pregnant or breastfeeding women
* Patients undergoing immediate breast reconstruction with Deep Inferior
* Epigastric Perforator (DIEP) o Transverse Rectus Abdominal Muscle techniques (TRAM) .
* Emergency procedures
* Documented allergy to chlorhexidine gluconate
* Antibiotic use in the fourteen days prior to surgical date
* Patients with a history or suspicion of breast cancer surgery outside the INCan in the previous three months.
* Patients who do not speak spanish, diagnosed with a psychiatric disorder and in whom a minimum follow-up of 14 days couldn't be feasible because of operative difficulties (eg.

place of residence or reference to other health institutions).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with drain bulb fluid bacterial colonization at the first and second week postoperative. | Approximately 1 or 2 weeks after surgery
  Bacterial growth was defined as plate growth >10*5 colony forming unit (CFU). Drains were removed at variable times across patients, per clinical indication. When clinically indicated, some patients did have their drains removed at the one week visit, in which case they only had one bulb fluid culture.
Number of subjects with drain tip bacterial colonization at removal. | Approximately at the second and/or third week after surgery
  Bacterial growth was defined as plate growth >15 CFU by semiquantitative technique or >10*5 CFU by sonication and fluid culture. Drains were removed at variable times across patients, per clinical indication.

SECONDARY OUTCOMES:
Number of Subjects With Surgical Site Infection Within 30 Days | Approximately 30 days after surgery
  Surgical site infection was diagnosed according the definitions given by the Centers for Disease Control and Prevention (CDC).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Results at the end of study

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Instituto Nacional de Geografía y estadística. "Estadísticas a propósito del día mundial de la lucha contra el cáncer de mama (19 de octubre)". Recuperado el 15 de febrero del 2016, de www.inegi.org.mx/aproposito/mama0
- [Background] Arce et al. Oncoguía: Cáncer de Mama. Cancerología 6, 2001; p77-86.
- [Background] Vilar-Compte D, Mohar A, Sandoval S, de la Rosa M, Gordillo P, Volkow P. Surgical site infections at the National Cancer Institute in Mexico: a case-control study. Am J Infect Control. 2000 Feb;28(1):14-20. doi: 10.1016/s0196-6553(00)90006-3. PMID 10679132
- [Background] Olsen MA, Chu-Ongsakul S, Brandt KE, Dietz JR, Mayfield J, Fraser VJ. Hospital-associated costs due to surgical site infection after breast surgery. Arch Surg. 2008 Jan;143(1):53-60; discussion 61. doi: 10.1001/archsurg.2007.11. PMID 18209153
- [Background] Olsen MA, Lefta M, Dietz JR, Brandt KE, Aft R, Matthews R, Mayfield J, Fraser VJ. Risk factors for surgical site infection after major breast operation. J Am Coll Surg. 2008 Sep;207(3):326-35. doi: 10.1016/j.jamcollsurg.2008.04.021. Epub 2008 Jun 26. PMID 18722936
- [Background] Edwards JR, Peterson KD, Mu Y, Banerjee S, Allen-Bridson K, Morrell G, Dudeck MA, Pollock DA, Horan TC. National Healthcare Safety Network (NHSN) report: data summary for 2006 through 2008, issued December 2009. Am J Infect Control. 2009 Dec;37(10):783-805. doi: 10.1016/j.ajic.2009.10.001. No abstract available. PMID 20004811
- [Background] Felippe WA, Werneck GL, Santoro-Lopes G. Surgical site infection among women discharged with a drain in situ after breast cancer surgery. World J Surg. 2007 Dec;31(12):2293-9; discussion 2300-1. doi: 10.1007/s00268-007-9248-3. PMID 17917771
- [Background] Ruvalcaba-Limon E, Robles-Vidal C, Poitevin-Chacon A, Chavez-Macgregor M, Gamboa-Vignolle C, Vilar-Compte D. Complications after breast cancer surgery in patients treated with concomitant preoperative chemoradiation: A case-control analysis. Breast Cancer Res Treat. 2006 Jan;95(2):147-52. doi: 10.1007/s10549-005-9058-y. Epub 2005 Dec 1. PMID 16319989
- [Background] Prospero E, Cavicchi A, Bacelli S, Barbadoro P, Tantucci L, D'Errico MM. Surveillance for surgical site infection after hospital discharge: a surgical procedure-specific perspective. Infect Control Hosp Epidemiol. 2006 Dec;27(12):1313-7. doi: 10.1086/509838. Epub 2006 Nov 21. PMID 17152028
- [Background] Vilar-Compte D, Jacquemin B, Robles-Vidal C, Volkow P. Surgical site infections in breast surgery: case-control study. World J Surg. 2004 Mar;28(3):242-6. doi: 10.1007/s00268-003-7193-3. Epub 2004 Feb 17. PMID 14961196
- [Background] Vilar-Compte D, Rosales S, Hernandez-Mello N, Maafs E, Volkow P. Surveillance, control, and prevention of surgical site infections in breast cancer surgery: a 5-year experience. Am J Infect Control. 2009 Oct;37(8):674-9. doi: 10.1016/j.ajic.2009.02.010. Epub 2009 Jun 24. PMID 19556033
- [Background] Vilar-Compte D, Roldan-Marin R, Robles-Vidal C, Volkow P. Surgical site infection (SSI) rates among patients who underwent mastectomy after the introduction of SSI prevention policies. Infect Control Hosp Epidemiol. 2006 Aug;27(8):829-34. doi: 10.1086/506395. Epub 2006 Jul 20. PMID 16874643
- [Background] Landes G, Harris PG, Lemaine V, Perreault I, Sampalis JS, Brutus JP, Lessard L, Dionyssopoulos A, Nikolis A. Prevention of surgical site infection and appropriateness of antibiotic prescribing habits in plastic surgery. J Plast Reconstr Aesthet Surg. 2008 Nov;61(11):1347-56. doi: 10.1016/j.bjps.2008.02.008. Epub 2008 Jun 16. PMID 18558522
- [Background] Throckmorton AD, Hoskin T, Boostrom SY, Boughey JC, Holifield AC, Stobbs MM, Baddour LM, Degnim AC. Complications associated with postoperative antibiotic prophylaxis after breast surgery. Am J Surg. 2009 Oct;198(4):553-6. doi: 10.1016/j.amjsurg.2009.06.003. PMID 19800467
- [Background] Hedrick TL, Smith PW, Gazoni LM, Sawyer RG. The appropriate use of antibiotics in surgery: a review of surgical infections. Curr Probl Surg. 2007 Oct;44(10):635-75. doi: 10.1067/j.cpsurg.2007.06.006. No abstract available. PMID 18021817
- [Background] XXXIII Congreso Nacional de la Asociación Mexicana de Infectología y Microbiología Clínica, A.C. León, Guanajuato; 14-17 de mayo de 2008.
- [Background] Throckmorton AD, Boughey JC, Boostrom SY, Holifield AC, Stobbs MM, Hoskin T, Baddour LM, Degnim AC. Postoperative prophylactic antibiotics and surgical site infection rates in breast surgery patients. Ann Surg Oncol. 2009 Sep;16(9):2464-9. doi: 10.1245/s10434-009-0542-1. Epub 2009 Jun 9. PMID 19506959
- [Background] Penel N, Yazdanpanah Y, Chauvet MP, Clisant S, Giard S, Neu JC, Lefebvre D, Fournier C, Bonneterre J. Prevention of surgical site infection after breast cancer surgery by targeted prophylaxis antibiotic in patients at high risk of surgical site infection. J Surg Oncol. 2007 Aug 1;96(2):124-9. doi: 10.1002/jso.20796. PMID 17443747
- [Background] Jones DJ, Bunn F, Bell-Syer SV. Prophylactic antibiotics to prevent surgical site infection after breast cancer surgery. Cochrane Database Syst Rev. 2014 Mar 9;(3):CD005360. doi: 10.1002/14651858.CD005360.pub4. PMID 24609957
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Purushotham AD, McLatchie E, Young D, George WD, Stallard S, Doughty J, Brown DC, Farish C, Walker A, Millar K, Murray G. Randomized clinical trial of no wound drains and early discharge in the treatment of women with breast cancer. Br J Surg. 2002 Mar;89(3):286-92. doi: 10.1046/j.0007-1323.2001.02031.x. PMID 11872051
- [Background] Barbadoro P, Marmorale C, Recanatini C, Mazzarini G, Pellegrini I, D'Errico MM, Prospero E; Drainages Collaborative Working Group. May the drain be a way in for microbes in surgical infections? Am J Infect Control. 2016 Mar 1;44(3):283-8. doi: 10.1016/j.ajic.2015.10.012. Epub 2015 Dec 21. PMID 26717874
- [Background] Simchen E, Rozin R, Wax Y. The Israeli Study of Surgical Infection of drains and the risk of wound infection in operations for hernia. Surg Gynecol Obstet. 1990 Apr;170(4):331-7. PMID 2181714
- [Background] Degnim AC, Scow JS, Hoskin TL, Miller JP, Loprinzi M, Boughey JC, Jakub JW, Throckmorton A, Patel R, Baddour LM. Randomized controlled trial to reduce bacterial colonization of surgical drains after breast and axillary operations. Ann Surg. 2013 Aug;258(2):240-7. doi: 10.1097/SLA.0b013e31828c0b85. PMID 23518704
- [Background] Degnim AC, Hoskin TL, Brahmbhatt RD, Warren-Peled A, Loprinzi M, Pavey ES, Boughey JC, Hieken TJ, Jacobson S, Lemaine V, Jakub JW, Irwin C, Foster RD, Sbitany H, Saint-Cyr M, Duralde E, Ramaker S, Chin R, Sieg M, Wildeman M, Scow JS, Patel R, Ballman K, Baddour LM, Esserman LJ. Randomized trial of drain antisepsis after mastectomy and immediate prosthetic breast reconstruction. Ann Surg Oncol. 2014 Oct;21(10):3240-8. doi: 10.1245/s10434-014-3918-9. Epub 2014 Aug 6. PMID 25096386
- [Background] Weichman KE, Clavin NW, Miller HC, McCarthy CM, Pusic AL, Mehrara BJ, Disa JJ. Does the use of biopatch devices at drain sites reduce perioperative infectious complications in patients undergoing immediate tissue expander breast reconstruction? Plast Reconstr Surg. 2015 Jan;135(1):9e-17e. doi: 10.1097/PRS.0000000000000810. PMID 25539357
- [Background] Sankar B, Ray P, Rai J. Suction drain tip culture in orthopaedic surgery: a prospective study of 214 clean operations. Int Orthop. 2004 Oct;28(5):311-4. doi: 10.1007/s00264-004-0561-2. Epub 2004 Aug 14. PMID 15316674
- [Background] Guembe M, Martin-Rabadan P, Cruces R, Perez Granda MJ, Bouza E. Sonicating multi-lumen sliced catheter tips after the roll-plate technique improves the detection of catheter colonization in adults. J Microbiol Methods. 2016 Mar;122:20-2. doi: 10.1016/j.mimet.2016.01.004. Epub 2016 Jan 14. PMID 26778418
- [Background] Jost GF, Wasner M, Taub E, Walti L, Mariani L, Trampuz A. Sonication of catheter tips for improved detection of microorganisms on external ventricular drains and ventriculo-peritoneal shunts. J Clin Neurosci. 2014 Apr;21(4):578-82. doi: 10.1016/j.jocn.2013.05.025. Epub 2013 Aug 14. PMID 24326253
- [Background] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Jun;35(6):605-27. doi: 10.1086/676022. PMID 24799638